CLINICAL TRIAL: NCT03918213
Title: Normative Metrics of High-Resolution Anorectal Manometry With the Use of Solid-State Catheter in a Healthy Russian Cohort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Collaborators: State Scientific Centre of Coloproctology, Russian Federation (Other Government); Federal Research Centre of Nutrition and Biotechnology (Unknown)
Responsible Party: Principal Investigator, Vasily Isakov, MD, PhD, Professor, AGAF, Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HRAM-HVSS
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Healthy Subjects
Keywords: high-resolution anorectal manometry; solid-state catheter; healthy population; Russian population

STUDY DESIGN:
Intervention Model Description: Normative values for the routine procedure of high-resolution anorectal manometry for Russian population has not been studied yet. Some factors allows to suggest that normative values may differ from those obtained in other countries. This pilot study is aimed to either support the null-hypothesis of the presence of the differences or decline it. It is expected to obtain primary data that could be used for further work and planning of the cohort studies. During the study, healthy volunteers are to be examined with a registered diagnostic tool (i.e. high-resolution anorectal manometry with solid-state catheter). This diagnostic procedure is not intended as one for routine examination, therefore the study type is "interventional", though no pharmacological intervention or surgery is planned. The estimated sample size sufficient to reach the power of 80%, and type 1 error 0.05 was obtained with single-sample t-test of Statistica10 (StatSoft, USA)
Masking Description: No masking is possible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- healthy subjects examined with solid-state catheter (Experimental): healthy subjects - subjects without signs of functional and organic anorectal pathology
  Interventions: Diagnostic Test: High-Resolution anorectal manometry with the use of solid-state catheter

INTERVENTIONS:
Diagnostic Test: High-Resolution anorectal manometry with the use of solid-state catheter — High resolution anorectal manometry with the use of solid-state catheter will be performed to eligible subjects willing to participate in the study
  Other Names: High-resolution anorectal manometry, solid-state catheter

SUMMARY:
High resolution anorectal manometry (HRAM) normative values are still need to be studied in different populations and with the use of different (solid-state and water-perfused) systems. No studies on HRAM normative values in a Russian population without signs of functional and organic anorectal pathology has been carried out yet.

DETAILED DESCRIPTION:
High-resolution anorectal manometry (HRAM) is a modern technique used to evaluate the function of the rectum and its sphincters. It is intended to measure the resting pressure in the anal canal, as well as pressure during voluntary contraction of the external anorectal sphincter and pelvic floor muscles and to evaluate reactions to the functional tests.

Several studies have been performed to evaluate normative metrics of anorectal manometry to the moment, but most of them enrolled patients living in the US and countries of the Western Europe. Nutritional patterns, ethnic composition of the population and other factors may cause the differences in the mormative values of HRAM in different populations. Current study is organized to evaluate normative metrics of HRAM in a Russian healthy cohort.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in this clinical trial, confirmed by signed informed consent form.
* Patients of both sexes, aged 18 to 65 years inclusive.
* Permanent residence in the Russian Federation (capable citizens of Russia on the basis of a passport of a citizen of the Russian Federation).
* Absence of rectal diseases, confirmed by the results of clinical and instrumental examinations
* Ability to follow the instructions when high-resolution anorectal manometry procedure is performed.

Exclusion Criteria:

* Known diseases of the rectum on the basis of clinical and / or instrumental examination, including presence of complaints to difficulties with defecations that require manual aids or use of laxatives;
* Surgical interventions on pelvic organs in history;
* History of organ transplantation except for corneal transplantation and eye lens replacement surgery;
* Oncology of any localization, with the exception of skin cancer in situ;
* Severe concomitant pathology of any organs and systems, which, in the opinion of the researcher, makes it impossible to carry out the procedure of high-resolution anorectal manometry or if the procedure may cause the risk of worsen the patient's condition;
* Absence of anamnestic, clinical and laboratory signs of alcohol abuse (abuse will be considered in case of the use of more than 30 g of pure alcohol per day by males and the use of more than 20 g of pure alcohol per day by females;
* Use of illegal drugs, including history;
* Use of concomitant medications that can affect the motor function of the colon (including, but not limited to: calcium channel blockers, metoclopramide, m-cholinolytics, domperidone, nitrates, tricyclic antidepressants, opiates, beta-blockers, beta-adrenomimetics, alcohol). The duration of the period of non-use of these drugs should provide sufficient time for the complete cessation of their pharmacological action, but not less than two half-life periods.
* Pregnancy and breast-feeding;
* Technical impossibility to insert the catheter due to the previously known or current poor tolerability of high-resolution anorectal manometry procedure or due to the presence of anatomical features that make it impossible to insert the catheter

Criteria of non-inclusion of the data to the analysis:

- Patients may choose to stop their participation in the study by withdrawal of their previously signed consent, that leads to the exclusion of their data from the analysis.

The researcher should be guided by the following criteria, however, he may at any time terminate the patient's participation in the study on the basis of his own clinical judgment.

Cancellation of participation in the study can be carried out on the basis of the following events:

* Lack of the possibility to insert water-perfused catheter during high-resolution anorectal manometry procedure due to anatomical features or psychological state of the patient.
* Incomplete high-resolution anorectal manometry procedure.
* Presence of adverse event(s) during high-resolution anorectal manometry procedure, causing the further procedure impossible.
* Obtaining incomplete recording of high-resolution anorectal manometry parameters for any reason.
* Identification of the conditions described in the section "exclusion criteria" during examination of the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2023-04-25 (Estimated); Study Completion 2024-04-25 (Estimated)

PRIMARY OUTCOMES:
Resting anorectal pressure obtained with the use of solid-state catheter for high-resolution anorectal manometry | 1 min
  Anorectal pressure at rest, mm Hg
Maximal squeeze pressure obtained with the use of solid-state catheter for high-resolution anorectal manometry | 5 sec
  Maximal pressure when a squeeze test is performed, mm Hg
Maximal pressure of endurance squeeze test performed with the use of solid-state catheter for high-resolution anorectal manometry | 30 seconds
  mean pressure during test, mm Hg
Push test pressure obtained with the use of solid-state catheter for high-resolution anorectal manometry | 5 seconds
  mean pressure during push test, mm Hg
Cough test | 5 seconds
  Cough test pressure maximal pressure, mmHg
Pressure of the first sensation obtained with the use of solid-state catheter for high-resolution anorectal manometry | 1 minute
  Pressure of the first sensation by the test of reservoir function of the rectum, mm Hg
Pressure of the urge to defecate obtained with the use of solid-state catheter for high-resolution anorectal manometry | 1 minute
  Pressure of the urge to defecate by the test of reservoir function of the rectum, mm Hg
Maximal tolerate volume pressure obtained with the use of solid-state catheter for high-resolution anorectal manometry | 1 minute
  Maximal tolerate volume (of baloon) pressure by the test of reservoir function of the rectum, ml
First pain sensation pressure obtained with the use of solid-state catheter for high-resolution anorectal manometry | 1 minute
  Appearance of pain sensation by the test of reservoir function of the rectum, mm Hg

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Morozov, MD, PhD, Principal Investigator — Fedreral Research Center of Nutrition and Biotechnology; Oksana Fomenko, MD, PhD, Principal Investigator — State Scientific Center of Coloproctology
Locations (2):
- Russia (2):
  - Gastroenterology and Hepatology, FRC Nutrition and Biotechnology, Moscow
  - State Scientific Center of Coloproctology, Moscow

IPD SHARING:
Plan to Share IPD: Yes
Depersonalized individual data may be shared upon the study completion
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5 years
Access Criteria: by request